CLINICAL TRIAL: NCT05203874
Title: Contribution of Multimodal Imaging in Early Neonatal Coarctation of Aorta: CT-COARCT-PED
Brief Title: Contribution of Multimodal Imaging in Early Coarctation
Acronym: CT-COARCT-PED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0734
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Aortic Coarctation; Congenital Heart Disease
Keywords: Multimodal imaging; Neonatal coarctation; Radiation protection
MeSH Terms: conditions — Aortic Coarctation; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CT-Coarct-PED study is a multicentred observational study aiming to describe the population of early coarctation during the last 10 years in South of France. The secondary objective is to assess the importance of cross-sectional imaging in the surgical management of aortic coarctation in the first year of life

DETAILED DESCRIPTION:
Coarctation of the aorta is one of the most common congenital heart diseases (5 to 8%). This heart disease can clinically result in two major clinical presentation: a neonatal form, early and potentially severe, which will require urgent care. And a later form, the discovery of which may be fortuitous. Even in it neonatal presentation, aortic coarctation will not occur during the pregnancy. But the performance of prenatal screening makes it possible to predict a "risk of coarctation" based on criteria that have been clarified with practice and time. (hypoplasia of the left cavities, isthmus / canal ratio etc.) Surgically, there are multiple techniques that will take into account the anatomy of the aortic arch and whether or not it is hypoplastic, the associated heart defects and the patient's characteristics. The choice of this surgical technique is one of the predominant elements of the future prognosis of this heart disease (recoarctation, arterial hypertension, etc.) It is in this context that the contribution of multimodal imaging (echocardiography, angiography CT scan and cardiac MRI), can be a determining element in the choice made by the surgeon of the aortic plastic surgery technique, by detailing the anatomical but also hemodynamic specificities Despite the lack of technical difficulty in performing a cardiac ultrasound in a newborn or an infant, the use of a cross sectional imaging (as CT angiography) is common in order to obtain a more comprehensive assessment of the aortic arch using 2D or 3D reconstruction techniques.

However, current practices in terms of radiation protection encourage us to limit the irradiation of our patients especially if the are to be expose potentially repeatedly to radiation during their medical care.

Thus, this multicenter study aims to clarify the role of cross-sectional imaging in the surgical management of aortic coarctation in the first year of life

ELIGIBILITY:
Inclusion criteria:

* Patients <1 years old
* Aortic coarctation in the first year of life
* Surgical management in one of the four participating centers
* No associated heart defect

Exclusion criteria

- age > 1 years

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all newborns who have had coarctation surgery during the first month of life in one of the four center included during the period between 2011 and 2021
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-29 (Estimated)

PRIMARY OUTCOMES:
Description of all cases of neonatal coarctations | day 1
  Description of all cases of neonatal coarctations in 4 surgical centers (Bordeaux Marseille, Nantes and Toulouse) over the years 2011 to 2021

SECONDARY OUTCOMES:
Level of agreement between the surgical procedure envisaged | day 1
  Level of agreement between the surgical procedure envisaged after a virtual staff
Level of agreement between the surgical procedure envisaged | day 1
  Level of agreement between the surgical procedure envisaged after the surgical procedure realized in real life

CONTACTS AND LOCATIONS:
Overall Officials: Oscar WERNER, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC